CLINICAL TRIAL: NCT05322161
Title: Yoga in the NICU for Parents (YiN): a Clinical Pilot Study
Brief Title: Yoga in the NICU for Parents Study
Acronym: YiN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Sara Neches, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00003325; SITE00001252 (Other: University of Washington)
Record Dates: First submitted 2022-03-03; First posted 2022-04-11 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Postpartum Depression; Anxiety; Depression; Stress Disorder; Prematurity
Keywords: yoga; meditation
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders; Depression; Stress Disorders, Traumatic; Premature Birth

STUDY DESIGN:
Intervention Model Description: Control group receives standard of care for parent support. Interventional group receives virtual yoga classes in addition to standard of care for parent support.
Who Masked: Investigator
Masking Description: Investigator is blinded to study allocation (yoga or control group) prior to enrollment. Once participant is randomized the investigator will know which group the participant is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Parents will experience usual care including all available parental support as practiced in the specific site NICU.
- Yoga Group (Experimental): In addition to usual care, the parents randomized to the intervention group will be provided a yoga mat and participate in 30-min online led yoga sessions done at least twice weekly at the parent's pace using a secure, virtual platform (website).
  Interventions: Behavioral: yoga classes

INTERVENTIONS:
Behavioral: yoga classes — There will be 6 total yoga classes (one introduced per week for a 6 week period). Each yoga session will be divided into three components, which will vary in duration based on a curriculum designed specifically with the post-partum state of mothers in mind:
  1. Yoga postures (Asana) = low impact gentle postures meant to be done individually
  2. Breathing techniques (Pranayama) = deliberate modifications of breath such as rapid diaphragmatic breathing, slow/deep breathing, alternate nostril breathing, breath holding
  3. Meditation (Dhyana) = guided meditation
  Arms: Yoga Group

SUMMARY:
The purpose of this proposal is to test the efficacy of yoga as a mind and body intervention to decrease stress, anxiety, and depression in parents of critically ill neonates hospitalized in the Seattle Children's and University of Washington neonatal intensive care units (NICUs).

DETAILED DESCRIPTION:
Preterm infants are often critically ill and require prolonged hospitalization in neonatal intensive care units (NICUs). The care of these infants is often regionalized so that specialized treatment can be performed in centers with specific expertise. An unintended consequence of regionalization of care is the physical and emotional isolation parents experience when a child is hospitalized far from family, friends, and work. As a result of these stressors, loss of parental control, autonomy, and concern for a child's wellbeing, nearly half of NICU mothers develop anxiety, depression, or posttraumatic stress disorder, and this may persist for years.

Helping parents cope with the birth and hospitalization of a preterm infant is critical for the parents' health and wellbeing, as well as for the optimal development of the child, as parental anxiety and depression may affect parent-child bonding and result in altered child development. The practice of yoga, which encompasses physical postures (asana), but also includes breathing techniques (pranayama), and meditation (dhyana), has proven benefits in many areas of medicine and wellness including stress management, mental and emotional health and promoting sleep. Given the positive effects on both physical and emotional health, these mind and body techniques are promising as a therapeutic modality by which parental stress, anxiety and depression could be reduced.

This study is unique in that previous studies of yoga have not occurred in hospital settings and have not included subjects in an acute state of distress such as parents of critically ill hospitalized neonates. Furthermore, in the current COVID-19 environment it is important to explore ways to make yoga interventions available to families by remote access, and to test whether this approach is successful.

This will be a randomized controlled pilot study to elucidate the optimal research strategy with which to implement mind and body interventions for parents of NICU patients, at two sites (University of Washington NICU and Seattle Children's Hospital NICU). We aim to enroll 40 NICU mothers and any of their interested partners in the study. We will approach parents after day 10 of infant admission to NICU and begin participation by day 14 of NICU admission.

The investigators hypothesize that a combined program of breath work, physical practice and meditation will decrease parental stress, anxiety, and depression in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* NICU inpatients born <32 weeks gestation at birth and/or <1500g, OR estimated length of stay ≥6 weeks
* Parents of current NICU inpatients born <32 weeks gestation at birth and/or <1500g OR estimated length of stay ≥6 weeks
* Parents with any level of experience with yoga (none to regular practitioner)
* Child has been admitted to the NICU for at least 10 days
* Parent age ≥18 years
* Parent speaks and reads in either English or Spanish

Exclusion Criteria:

* Expected length of stay of NICU inpatient <6 weeks
* Parent does not speak or read in English only speaks or reads in a language other than English or Spanish
* Parent plans to relinquish child
* Child or parents are too unstable as assessed by the Attending Physician

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change in parental depression, anxiety and stress score over time | Administered at three time points: At randomization, after 3-weeks in the study, after 6-weeks at the conclusion of the study
  The depression, anxiety & stress scale (DASS-21) is validated in English and Spanish and is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three sub scales (depression, anxiety and stress) contain 7 questions with answers valued on a scale of 0-3. Scores for depression, anxiety, and stress are calculated by summing the scores for the relevant items. Each sub scale score is multiplied by 2 and totaled to generate a DASS 21 score. Analysis will include mean/SD and median of total score and comparison of median DASS 21 score between pre and post-intervention. A high score on the DASS 21 means worse depression, anxiety and stress.
Measure of NICU parent stress | Administered at three time points: At randomization, after 3-weeks in the study, after 6-weeks at the conclusion of the study
  The Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU) is a 26-item self-report scale designed to measure the degree of stress experienced by parents during hospitalization. This scale has been validated in multiple languages including English and Spanish. Analysis will assess parents' overall level of stress engendered by the NICU environment. All individuals receive a score on each item, with those not having the experience (e.g N/A) receiving a "1" indicating no stress was experienced. Score will be generated by a total sum of: sub scale 1: Sights and Sounds (sum/5)+ sub scale 2: Infant behavior and appearance (sum/14)+ sub scale 3: Parental Role Alteration (sum/7). Analysis to include: mean/SD for each sub scale and mean/SD for total score for each participant. Mean scores on the PSS:NICU will be compared across the three time-points and between parents in each arm (intervention and control). A higher score on the PSS:NICU means higher NICU parent stress.
Measure of parent-child bonding | Once after 6-weeks at the conclusion of the study
  Postpartum Bonding Questionnaire (PBQ) was developed to detect mother-infant bonding disturbances in the postnatal period. Participants rate how often they agree with statements on a 6-point Likert scale ranging from always (score 0) to never (score 5) with low scores denoting good bonding. We plan to use 2 of the four sub scales (19-item self-report scale). A score of >/= 12 on scale 1 and >/= 13 on scale 2 indicates worse parent-child bonding.

SECONDARY OUTCOMES:
Infant Length of Stay | From date of admission until infant discharge home or transfer to another institution, up to a maximum of 32 weeks.
  Length of stay (days) from admission to discharge home or transfer to other institution, as documented on the discharge or transfer summary.
Length of assisted ventilation (days) | From date of admission through discharge home or transfer to another institution, up to a maximum of 32 weeks.
  Length of time (days) that infant required either invasive or non-invasive ventilation, as documented on the discharge or transfer summary.
Breastfeeding at discharge | At the date of discharge to home, up to a maximum of 32 weeks.
  Documentation of whether infant is doing any breastfeeding at discharge (yes/no) as documented on the discharge summary.
Yoga class participation | From randomization through the conclusion of the 6-week study period
  Participation in the yoga intervention will be tracked on the study website to assess number of sessions started (n)
Duration of participation in yoga classes | From randomization through the conclusion of the 6-week study period
  Participation in the yoga intervention will be tracked on the study website to assess duration of participation (minutes).
Postpartum Depression | Up to 4 weeks after admission
  The Edinburgh Postnatal Depression Scale (EPDS) has been validated in both women and men, and consists of 10 questions. The total score is determined by adding together the scores for each of the 10 items. Cut-off scores ranged from 9 to13 points with higher scores indicating worse post-partum depression. EPDS is administered to mothers by the NICU social worker between day 10-14 of admission. Participating fathers will fill out an EPDS survey as part of enrollment in this study.
Parent Satisfaction with Yoga Intervention | Once after 6-weeks at the conclusion of the study
  Course completion study filled out by all participants at the conclusion of the study. There will be specific questions geared to the intervention group to qualitatively assess parent satisfaction with the yoga intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Neches, MD, Principal Investigator — Seattle Children's Hospital
Locations (2):
- United States (2):
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported after de-identification (texts, tables, figures and appendices). Study protocol, statistical analysis plan and analytic code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: beginning 3 months and ending 5 years following the article publication
Access Criteria: Proposals should be directed to skneches@uw.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Treyvaud K, Spittle A, Anderson PJ, O'Brien K. A multilayered approach is needed in the NICU to support parents after the preterm birth of their infant. Early Hum Dev. 2019 Dec;139:104838. doi: 10.1016/j.earlhumdev.2019.104838. Epub 2019 Aug 27. PMID 31471000
- [Background] Yaari M, Treyvaud K, Lee KJ, Doyle LW, Anderson PJ. Preterm Birth and Maternal Mental Health: Longitudinal Trajectories and Predictors. J Pediatr Psychol. 2019 Jul 1;44(6):736-747. doi: 10.1093/jpepsy/jsz019. PMID 30977828
- [Background] Pace CC, Spittle AJ, Molesworth CM, Lee KJ, Northam EA, Cheong JL, Davis PG, Doyle LW, Treyvaud K, Anderson PJ. Evolution of Depression and Anxiety Symptoms in Parents of Very Preterm Infants During the Newborn Period. JAMA Pediatr. 2016 Sep 1;170(9):863-70. doi: 10.1001/jamapediatrics.2016.0810. PMID 27428766
- [Background] Winter L, Colditz PB, Sanders MR, Boyd RN, Pritchard M, Gray PH, Whittingham K, Forrest K, Leeks R, Webb L, Marquart L, Taylor K, Macey J. Depression, posttraumatic stress and relationship distress in parents of very preterm infants. Arch Womens Ment Health. 2018 Aug;21(4):445-451. doi: 10.1007/s00737-018-0821-6. Epub 2018 Mar 3. PMID 29502280
- [Background] Moehler E, Brunner R, Wiebel A, Reck C, Resch F. Maternal depressive symptoms in the postnatal period are associated with long-term impairment of mother-child bonding. Arch Womens Ment Health. 2006 Sep;9(5):273-8. doi: 10.1007/s00737-006-0149-5. Epub 2006 Sep 8. PMID 16937313
- [Background] Treyvaud K, Anderson VA, Lee KJ, Woodward LJ, Newnham C, Inder TE, Doyle LW, Anderson PJ. Parental mental health and early social-emotional development of children born very preterm. J Pediatr Psychol. 2010 Aug;35(7):768-77. doi: 10.1093/jpepsy/jsp109. Epub 2009 Dec 2. PMID 19955253
- [Background] Treyvaud K, Anderson VA, Howard K, Bear M, Hunt RW, Doyle LW, Inder TE, Woodward L, Anderson PJ. Parenting behavior is associated with the early neurobehavioral development of very preterm children. Pediatrics. 2009 Feb;123(2):555-61. doi: 10.1542/peds.2008-0477. PMID 19171622
- [Background] Kerstis B, Aarts C, Tillman C, Persson H, Engstrom G, Edlund B, Ohrvik J, Sylven S, Skalkidou A. Association between parental depressive symptoms and impaired bonding with the infant. Arch Womens Ment Health. 2016 Feb;19(1):87-94. doi: 10.1007/s00737-015-0522-3. Epub 2015 Apr 10. PMID 25854998
- [Background] de Cock ESA, Henrichs J, Klimstra TA, Janneke B M Maas A, Vreeswijk CMJM, Meeus WHJ, van Bakel HJA. Longitudinal Associations Between Parental Bonding, Parenting Stress, and Executive Functioning in Toddlerhood. J Child Fam Stud. 2017;26(6):1723-1733. doi: 10.1007/s10826-017-0679-7. Epub 2017 Feb 27. PMID 28572718
- [Background] Trkulja V, Baric H. Current Research on Complementary and Alternative Medicine (CAM) in the Treatment of Anxiety Disorders: An Evidence-Based Review. Adv Exp Med Biol. 2020;1191:415-449. doi: 10.1007/978-981-32-9705-0_22. PMID 32002940
- [Background] Cramer H, Lauche R, Anheyer D, Pilkington K, de Manincor M, Dobos G, Ward L. Yoga for anxiety: A systematic review and meta-analysis of randomized controlled trials. Depress Anxiety. 2018 Sep;35(9):830-843. doi: 10.1002/da.22762. Epub 2018 Apr 26. PMID 29697885
- [Background] Cramer H, Anheyer D, Saha FJ, Dobos G. Yoga for posttraumatic stress disorder - a systematic review and meta-analysis. BMC Psychiatry. 2018 Mar 22;18(1):72. doi: 10.1186/s12888-018-1650-x. PMID 29566652
- [Background] Cramer H, Anheyer D, Lauche R, Dobos G. A systematic review of yoga for major depressive disorder. J Affect Disord. 2017 Apr 15;213:70-77. doi: 10.1016/j.jad.2017.02.006. Epub 2017 Feb 7. PMID 28192737
- [Background] Brockington IF, Fraser C, Wilson D. The Postpartum Bonding Questionnaire: a validation. Arch Womens Ment Health. 2006 Sep;9(5):233-42. doi: 10.1007/s00737-006-0132-1. Epub 2006 May 4. PMID 16673041
- [Background] Matthey S, Barnett B, Kavanagh DJ, Howie P. Validation of the Edinburgh Postnatal Depression Scale for men, and comparison of item endorsement with their partners. J Affect Disord. 2001 May;64(2-3):175-84. doi: 10.1016/s0165-0327(00)00236-6. PMID 11313084

DOCUMENTS (1):
  • Study Protocol (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT05322161/Prot_000.pdf